CLINICAL TRIAL: NCT06107764
Title: Cerebellar Modulation of Cognition in Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Eve Lewandowski, Associate Professor of Psychiatry, McLean Hospital, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2023P002474
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder I; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study design is a crossover design i.e. all participants will receive all three rTMS interventions (iTBS, cTBS, sham rTMS). The participant will be blinded to which intervention is happening on a given study visit. The order of these visits will be determined randomly for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Intermittent theta burst stimulation (iTBS) (Active Comparator): Participants complete MRI scanning and cognitive testing followed by rTMS (iTBS pattern) followed by repeat cognitive testing and MRI scanning
  Interventions: Device: intermittant theta burst stimulation (iTBS)
- continuous theta burst stimulation (cTBS) (Active Comparator): Participants complete MRI scanning and cognitive testing followed by rTMS (cTBS pattern) followed by repeat cognitive testing and MRI scanning
  Interventions: Device: continuous theta burst stimulation (cTBS)
- sham rTMS (Sham Comparator): Participants complete MRI scanning and cognitive testing followed by sham rTMS followed by repeat cognitive testing and MRI scanning
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: intermittant theta burst stimulation (iTBS) — iTBS consists of 2 s trains of 3 pulses at 50 Hz, repeated at 5 Hz, every 10s for a total of 600 pulses.
  Arms: Intermittent theta burst stimulation (iTBS)
Device: continuous theta burst stimulation (cTBS) — cTBS consists of 3 pulses at 50 Hz repeated at 5 Hz (every 200ms) continuously for a total of 600 pulses
  Arms: continuous theta burst stimulation (cTBS)
Device: sham rTMS — sham rTMS does not deliver a significant change in magnetic field strength
  Arms: sham rTMS

SUMMARY:
The goal of this clinical trial is to learn about cognition in psychotic disorders (schizophrenia, bipolar disorder, and schizoaffective disorder). The main question it aims to answer is: Can we use magnetic stimulation to change processing speed (how quickly people can solve challenging tasks).

Participants will be asked to perform cognitive tasks (problem-solving) and undergo brain scans before and after transcranial magnetic stimulation (TMS). TMS is a way to non-invasively change brain activity. Forms of TMS are FDA-approved to treat depression and obsessive compulsive disorder. In this study, we will use a different form of TMS to temporarily change brain activity to observe how that changes speed in problem-solving.

DETAILED DESCRIPTION:
Psychotic disorders including schizophrenia, bipolar disorder, and related illnesses are severe, debilitating, and often fatal. Cognitive impairments in psychosis are among the leading predictors of disability and poor quality of life; despite this, there are no first-line interventions to target these symptoms.

This trial will test the hypothesis that cognitive performance in these disorders is modifiable and specifically that it can be modified non-invasively. Transcranial magnetic stimulation (TMS) is a neuromodulation technique that utilizes magnets to alter brain activity non-invasively. TMS has received FDA approval as a therapeutic intervention for multiple psychiatric disorders. In this study, we will use different forms of TMS to modulate a specific brain circuit and we will measure the outcomes of this circuit manipulation. These outcomes include performance on cognitive tests and also changes to the circuit itself that we can measure using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years
* Diagnosis of a psychotic disorder (i.e. schizophrenia or schizoaffective disorder or bipolar disorder type I)
* Must be able to read, speak and understand English
* Must be judged by study staff to be capable of completing the study procedures
* Participants will be in stable outpatient treatment with no recent (within the past 30 days) hospitalizations or changes in their medication regimens.

Exclusion Criteria:

* Diagnostic and Statistical Manual 5 diagnosis of moderate substance use disorder within the past month
* Conditions that might result in increased risks of side effects or complications from rTMS or MRI, including:

  * Intracranial pathology from a known genetic disorder (e.g., Neurofibromatosis 1, tuberous sclerosis) or from acquired neurologic disease (e.g. stroke, tumor), cerebral palsy, history of severe head injury, or significant dysmorphology;
  * History of fainting spells of unknown or undetermined etiology that might constitute seizures
  * History of multiple seizures or diagnosis of epilepsy
  * Any progressive (e.g., neurodegenerative) neurological disorder such as multiple sclerosis or Parkinson's disease
  * Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
  * Metal implants (excluding dental fillings) unless cleared by the responsible covering MD (i.e. MRI compatible joint replacement)
  * Pacemaker
  * Implanted medication pump
  * Vagal nerve stimulator
  * Deep brain stimulator or transcutaneous electric nerve stimulation unit
  * Ventriculo-peritoneal shunt
  * Signs of increased intracranial pressure
  * Intracranial lesion
  * History of head injury resulting in prolonged loss of consciousness (>15minutes) or neurological sequelae
  * Pregnancy: All participants capable of becoming pregnant will be required to have a pregnancy test; any participant who is pregnant will not be enrolled in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
BACS Symbol Coding test | eight minutes before TMS and one minute after TMS on each of the three TMS visit days
  The BACS Symbol coding test is a test of information processing speed
BACS Digit Sequence test | five minutes before TMS and four minutes after TMS on each of the three TMS visit days
  The BACS digit sequence test is a test of working memory performance
functional Magnetic Resonance Imaging | fifteen minutes before TMS and nine minutes after TMS on each of the three TMS visit days
  resting-state (task free) functional connectivity

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No